CLINICAL TRIAL: NCT02350894
Title: Microstructural Changes in the Brain During Recovery After Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Hammel Neurocenter (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-139-14
Record Dates: First submitted 2015-01-19; First posted 2015-01-30 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2016-10

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- mTBI subjects: mTBI subjects with ongoing symptoms
  Interventions: Behavioral: Graded and behavevial theraphy

INTERVENTIONS:
Behavioral: Graded and behavevial theraphy — Graded and behavevial theraphy

SUMMARY:
This study examines the possible microstructural changes in the brain during recovery after mTBI using diffusion MRI.

DETAILED DESCRIPTION:
This study is embedded in a larger randomized controlled trial (RCT) (ClinicalTrials.gov ID: NCT02337101) from which the subjects are recruited and will separately examine the possible microstructural changes in the brain during recovery after mild traumatic brain injury (mTBI) in subjects with ongoing symptoms more than 2 month after mTBI in both groups from the RCT.

Several biomarkers and brain areas has been investigated as possible sites of injury after mTBI. The nature of the diffuse chronic post-concussion symptoms (PCS) makes corpus callosum (CC), thalamus (THA) and hippocampus (HIP) interesting because of their central position and connection to widespread motor, sensory and cognitive processes and other brain areas. In most prior studies conventional magnetic resonance imaging (MRI) has failed to detect pathology especially in the chronic phase after mTBI. Diffusional Kurtosis Imaging (DKI) and Diffusional Tensor Imaging (DTI) are more sensitive to microstructural changes and might serve as biomarkers in the brain after mTBI.

We hypothesized that a change in symptoms (as measured by cognitive performance and self reported symptoms) will correlate with a change in microstructural changes (as measured with DKI) in thalamus, corpus callosum and hippocampus from baseline 2-6 month after mTBI to follow up 6 month after.

Separate correlations will also be made for both treatment and control group within the cohort.

ELIGIBILITY:
Inclusion Criteria:

* Concussion caused by a head trauma according to the diagnostic criteria recommended by the Danish Consensus Report on Commotio Cerebri within the last 2-6 months. The criteria are based on recommendations by the WHO Task Force, but with the amendment, that there must have been a direct contact between the head and an object in order to rule out pure acceleration - deceleration traumas.
* Age 18 to 30 years at the time of the head trauma.
* Able to understand, speak and read Danish.
* Patients with symptoms on at least three items on the Rivermead Post Concussion Symptoms Questionnaire (RPQ) rated as moderate or severe problem. PCS have to be subjectively rated as causing substantial impairment in daily life.
* Suitable for MRI examination

Exclusion Criteria:

* Objective neurological findings from neurological examination and / or acute trauma CT scan, indicating other neurological diseases or brain damage.
* Previous concussion leading to persistent PCS within the last two years.
* Severe abuse of alcohol, prescription drugs and / or illegal drugs.
* Psychiatric morbidity or severe neurological disease that impedes participation in the treatment, i.e. Bipolar Disorder, autism, psychotic disorder (lifetime), multiple sclerosis etc.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Mild traumatic brain injury subjects with ongoing symptoms 2-6 months after trauma
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Microstructural changes in the thalamus, corpus callosum and hippocampus between baseline and follow up, as measured by Diffusion kurtosis imaging (DKI) | Baseline 2-6 month after mTBI with follow up 6 month after
  MRI measurement

SECONDARY OUTCOMES:
Microstructural changes in the thalamus, corpus callosum and hippocampus from baseline to follow up, as measured by Diffusion tensor imaging (DTI) | Baseline 2-6 month after mTBI with follow up 6 month after
  MRI measurement
Change in post-concussion symptoms from baseline to follow up, as measured by Rivermead post-concussion questionnaire (RPQ) and headache (VAS scale) | Baseline 2-6 month after mTBI with follow up 6 month after
  Symptom score
Change in Cognitive performance from baseline to follow up, as measured by executive function, verbal and visual memory, processing speed, working memory, Visuospatial perception and construction | Baseline 2-6 month after mTBI with follow up 6 month after
  Cognitive test battery

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen F Nielsen, Professor, Principal Investigator — Hammel Neurocenter - Universitetsklinik for Neurorehabilitering, Aarhus Universi
Locations (1):
- Region Hospital Hammel Neurocenter, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trillingsgaard Naess-Schmidt E, Udby Blicher J, Moller Thastum M, Ulrikka Rask C, Wulff Svendsen S, Schroder A, Hogh Tuborgh A, Ostergaard L, Sangill R, Lund T, Norhoj Jespersen S, Roer Pedersen A, Hansen B, Fristed Eskildsen S, Feldbaek Nielsen J. Microstructural changes in the brain after long-term post-concussion symptoms: A randomized trial. J Neurosci Res. 2021 Mar;99(3):872-886. doi: 10.1002/jnr.24773. Epub 2020 Dec 15. PMID 33319932
- See also: The Research Clinic for Functional Disorders and Psychosomatics, Aarhus University Hospital — http://funktionellelidelser.dk/
- See also: Center of Functionally Integrative Neuroscience, Aarhus University, Aarhus University Hospital — http://cfin.au.dk/